CLINICAL TRIAL: NCT06337162
Title: A Pilot Study of Neoadjuvant INCB099280 in Patients With Hepatocellular Carcinoma Awaiting Liver Transplant
Brief Title: Pre-Transplant INCBB099280 for Hepatocellular Carcinoma (HCC)
Acronym: HCC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Incyte made a strategic business decision to stop enrollment to all ongoing oral PD-L1 (99280) studies. This decision was made based on an internal review and reprioritization of the existing pipeline.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 20223; IRB#855195 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB099280 (Experimental): Study participants will receive the recommended phase II dose (400mg/kg) of INCB099280 orally on days 1 through 28 of each 28-day cycle until liver transplant.
  Interventions: Drug: INCB099280

INTERVENTIONS:
Drug: INCB099280 — 400 mg Tablet

SUMMARY:
This is a pilot safety study of the oral PD-L1 inhibitor INCB099280 in patients with HCC awaiting liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Must have hepatocellular carcinoma (HCC) that is within criteria for liver transplantation per review at multidisciplinary tumor board. This includes HCC tumors meeting downstaging criteria, per United Network for Organ Sharing (UNOS) guidelines.
* Age > 18 years and ability to understand and the willingness to sign a written informed consent document.
* No prior systemic therapies for HCC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Child-Pugh cirrhosis score of A5, A6, or B7
* Must be willing to comply with protocol procedures.
* Patients who are undergoing locoregional therapies must have resolution of clinical (i.e. not laboratory) adverse effects associated with the locoregional therapy to grade ≤1 or baseline (whichever is higher).
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days of the first dose of INCB099280.
* Must have adequate organ and hematopoietic function within 7 days of initiation of study therapy (including Cycle 1 Day 1 labs if needed).

Exclusion Criteria:

* Any history of a serious medical or psychiatric condition that would prevent the subject from signing the informed consent form.
* Intercurrent illness that might interfere with compliance or study completion.
* Pregnant, expecting to conceive, or breastfeeding starting with the screening visit through 190 days after the last dose of study treatment or expecting to father children starting with the screening visit through 100 days after the last dose of study treatment.
* Subjects may not receive concomitant anticancer agents (except protocol specified INCB099280). Long-term hormonal agents used in the adjuvant setting for other cancers (e.g. tamoxifen for breast cancer, leuprolide for prostate cancer) are permitted.
* Uncontrolled ascites (i.e. requiring paracentesis).
* Hepatic encephalopathy symptoms within 6 months prior to starting study therapy.
* Portal vein invasion or extrahepatic metastatic disease.
* Treatment with non-steroidal systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment. Systemic agents for skin-only conditions such as atopic dermatitis or psoriasis may be permissible at the discretion of the Principal Investigator.
* Any concurrent condition requiring the continued or anticipated use of systemic steroids beyond physiologic replacement dosing (excluding non-systemic inhaled, topical skin, nasal, and/or ophthalmic corticosteroids). All other systemic corticosteroids above physiologic replacement dosing must be discontinued at least 2 weeks prior to first study treatment. Patients who receive a corticosteroid pulse for IV contrast allergies are eligible.
* Active drug or alcohol use or dependence as documented in the chart that, in the opinion of the investigator, would interfere with adherence to study requirements or interfere with eligibility for liver transplantation.
* Serious active bacterial or fungal infection requiring oral or intravenous antibiotics or antifungals at the start of protocol treatment. Participants may enroll after a 28-day washout period. Prophylactic or suppressive antibiotics (e.g. for spontaneous bacterial peritonitis prophylaxis, dental procedures, or surgical prophylaxis) are allowed.
* A second primary malignancy that, in the judgment of the investigator, may affect the interpretation of results and/or eligibility for liver transplantation. Exceptions may be made if the participant has undergone potentially curative therapy with no evidence of disease recurrence for 3 years since initiation of that therapy and the participant is otherwise a candidate for Liver Transplant (Note: The time requirement for no evidence of disease for 3 years does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, other noninvasive or indolent malignancies, or other in situ cancers if the presence or history of these cancers would not otherwise affect candidacy for liver transplant (LT)).
* Prior organ allograft or allogeneic bone marrow transplantation.
* Active autoimmune disease, except for vitiligo, type 1 diabetes mellitus, asthma, atopic dermatitis, psoriasis, or endocrinopathies manageable by hormone replacement; other autoimmune conditions with low risk of complications due to Immune Checkpoint Inhibitors (ICI) use may be allowable at the discretion of the Principal Investigator.
* Any other conditions judged by the investigator that would limit the evaluation of the subject.
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* If Hepatitis B surface antigen positive, must be on hepatitis B antiviral therapy for at least 21 days prior to starting study therapy and continue antiviral therapy for at least one year following cessation of study therapy.
* Impaired cardiac function or clinically significant cardiac disease: New York Heart Association Class III or IV cardiac disease, including preexisting clinically significant ventricular arrhythmia, congestive heart failure, or cardiomyopathy, unstable angina pectoris, acute myocardial infarction ≤ 6 months before study participation, other clinically significant heart disease (ie, uncontrolled ≥ Grade 3 hypertension), and/or Clinically significant ECG abnormality, including Corrected QT Interval Using Fridericia's Formula (QTcF) interval > 480 milliseconds (Note: If a single ECG tracing at screening is > 480 milliseconds, the average of a triplicate ECG may be used).
* History or evidence of interstitial lung disease, including noninfectious pneumonitis.
* Presence of gastrointestinal conditions that may affect drug absorption, as well as those that interfere with gastrointestinal transit, including gastric bypass surgery, gastric sleeve, or gastric band.
* Diagnosis of primary immunodeficiency.
* HIV infection and any one or more of the following: Cluster of Differentiation 4 (CD4) + T-cell count < 200 cells/μL, detectable viral load, or antiretroviral therapy regimen containing moderate or potent CYP3A4/CYP3A5 inhibitors or inducers (Note: Participants modifying their HIV regimen to include only drugs without CYP3A4/5 inhibitors or inducers must be on a stable regimen for > 28 days prior to enrollment)
* Known hypersensitivity or severe reaction to any component of study drug or formulation components.
* Postoperative complications preventing the participant from adhering to protocol assessments and procedures.
* Received a live vaccine within 28 days of the planned start of study drug. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chickenpox, some shingles, yellow fever, rabies, Bacille Calmette-Guérin (BCG), and typhoid vaccines. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live-attenuated vaccines and are not allowed.
* Treatment with moderate and potent CYP3A4/CYP3A5 inhibitors or inducers Note: A washout period ≥ 10 days before the first dose of INCB099280 is required for prior treatment with CYP3A4/CYP3A5 inhibitors/inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Acute Cellular Rejection of Liver Transplant Attributed to Study Therapy | From liver transplant until 1 month after liver transplant
  Proportion of patients who undergo liver transplant who experience biopsy-proven acute cellular rejection of liver transplant using Banff Criteria within 1 month of liver transplantation that is at least possibly related to study therapy

SECONDARY OUTCOMES:
Acute Cellular Rejection of Liver Transplant Within 3 Months | From liver transplant until 3 months after liver transplant
  Proportion of patients who undergo liver transplant who experience biopsy-proven acute cellular rejection of liver transplant using Banff Criteria within 3 month of liver transplantation
Acute Cellular Rejection of Liver Transplant Within 1 Year | From liver transplant until 1 year after liver transplant
  Proportion of patients who undergo liver transplant who experience biopsy-proven acute cellular rejection of liver transplant using Banff Criteria within 1 year of liver transplantation
Toxicity Rates by Category and Grade | From start of study therapy to 1 month after liver transplant
  Treatment-emergent adverse events graded using CTCAE v. 5.0
Proportion of Patients Downstaged | From start of study therapy to liver transplant, an average of 6 months
  Proportion of patients outside of the Milan Criteria at study entry who undergo liver transplant
Pathologic Complete Response Rate | At time of liver transplant, an average of 6 months
  Proportion of patients undergoing liver transplant with a complete pathologic response on liver explant
Recurrence-Free Survival at 1 Year After Transplant | From liver transplant until 1 year after liver transplant
  Proportion of patients who undergo liver transplant without recurrence of hepatocellular carcinoma within 1 year after transplant
Overall Survival at 1 Year After Transplant | From liver transplant until 1 year after liver transplant
  Proportion of patients who undergo liver transplant who are alive 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karasic, MD, Principal Investigator — Abramson Cancer Center at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No